CLINICAL TRIAL: NCT06785259
Title: Complex Systems Analysis of the Impact of Mindfulness Intervention on Emotional Distress: A Study of Daily Interventions and Daily Diary
Brief Title: Mindfulness Interventions and Emotional Distress: A Daily Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E20250107
Record Dates: First submitted 2025-01-07; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIED group (Experimental): Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge, and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression, and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress(MIED) — Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.

SUMMARY:
This study hopes to explore whether the changes in rumination exhibited in Daily Diary mediates the effects of mindfulness intervention on alleviating emotional distress

DETAILED DESCRIPTION:
This study will employ a daily diary research design to collect detailed time-series data, capturing the dynamic evolution of participants' emotional changes. This approach not only facilitates the provision of robust evidence regarding the effects of mindfulness interventions but also offers valuable insights for refining and personalizing future intervention strategies.

Mindfulness involves observing one's current state of mind with an open, non-judgmental attitude, including awareness of breathing, bodily sensations, and actions (Wielgosz et al., 2019). With the widespread use of the internet and smartphones, there has been a rapid increase in the demand for mental health services, leading to the emergence of lightweight online mindfulness intervention programs that have garnered increasing attention (Taylor et al., 2021).

Mindfulness-based interventions (MBIs) can positively impact various aspects of individuals' lives (Wielgosz et al., 2019), including physical and mental health, cognitive abilities, emotions, and interpersonal relationships. Regular mindfulness training often leads to healthier behaviors, such as reduced substance abuse, decreased self-harm and suicidal behaviors, and alleviation of eating disorder symptoms (Schuman-Olivier et al., 2020). MBIs are applicable to both clinical and non-clinical populations: they benefit not only patients with physical or mental illnesses (Carlson, 2012; Turgon et al., 2019) but also those experiencing behavioral or emotional distress (Ju, 2022; Ma et al., 2018).

In addition to studying the efficacy of interventions, it is crucial to explore their mechanisms of action. Traditional methods of mechanism research have provided some evidence, defining mechanisms as "processes responsible for change," while mediators are "statistical explanations of the relationship between independent and dependent variables" (Kazdin, 2007, p.3). Currently, researchers have begun to investigate the mechanisms underlying mindfulness-based stress reduction (MBSR) and mindfulness-based cognitive therapy (MBCT) (Batink et al., 2013; Geschwind et al., 2011; Alsubaie et al., 2017).

However, traditional theoretical frameworks and analytical methods cannot adequately explain or capture sudden, nonlinear changes during the intervention process. Such phenomena can be better understood through complex systems theory. By applying complex network theory and methods, we can gain new insights into the complexity and dynamics of changes during the intervention process, identify intervention targets, uncover potential core targets, predict abrupt changes, and provide evidence for optimizing intervention targets and timing, thereby enhancing the effectiveness of intervention programs. Complex systems theory holds great promise for understanding the mechanisms of psychological interventions, yet few studies have examined the complex and dynamic changes in psychological variables during interventions from this perspective in the field of mindfulness research.

Therefore, in this study, we will first focus on several potential mechanism variables, specifically rumination, using the framework and analytical tools of complex systems theory to examine the complexity and dynamics of changes during online mindfulness interventions.

An increasing number of researchers are beginning to view rumination as a transdiagnostic pathological process closely related to the development and maintenance of various emotional disturbances (Ehring & Watkins, 2008; Nolen-Hoeksema & Watkins, 2011; Watkins & Roberts, 2020). Rumination is associated with multiple emotional disorders and their comorbid conditions, including depressive disorders and anxiety disorders (Nolen-Hoeksema, 2000; Nolen-Hoeksema, Wisco, & Lyubomirsky, 2008). Rumination is a negative thought pattern characterized by repetitive negative thinking about problems, the causes, meanings, and consequences of distress (Watkins, 2008). It typically involves negative self-evaluations and is considered a maladaptive emotion regulation strategy linked to reduced well-being (Brans et al., 2013).

In summary, most current mechanism studies have not rigorously characterized the processes underlying mindfulness interventions using multiple measurement points and appropriate statistical methods, nor have they simultaneously examined the complexity and dynamics of multiple mechanism variables and outcome variables in mindfulness interventions. Therefore, conducting daily diary research will provide valuable evidence for a deeper and more comprehensive understanding of how interventions work.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet.
* Subjects with insufficient Chinese ability.
* Subjects who have participated in mindfulness-based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week.
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder.
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-18 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Daily changes of mindfulness | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  The Daily Mindfulness Response Scale measures the frequency with which one returns to a nonjudgmental and unconditionally receptive present moment awareness during the day. Each item is rated on a scale ranging from 1 (rarely)to10(often). scores range from 4 to 40, with higher scores indicating higher levels of mindful responding
Daily changes of rumination | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  measured by Momentary repetitive negative thinking, night items, scores range from 9 to 63, with higher scores indicating higher levels of reprtitive negative thinking.
Daily changes of positive and negative affect | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily positive and negative affect were measured using the 10-itemInternational Positive and Negative Affect Schedule-Short Form Scale. Scores range from 5 to 25, with higher scores indicating higher levels of positive/negative affect.
Daily changes of emotional distress | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
daily changes of anxiety | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily Anxiety Severity and Impairment Scale,5 items, scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
daily changes of depression | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily Depression Severity and Impairment Scale,5 items, scores range from 0 to 20, with higher scores indicating higher levels of depression.
Daily changes of the Brief State Rumination Inventory | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  he Brief State Rumination Inventory comprises eight items designed to measure an individual's state rumination tendency at a given moment, encompassing aspects such as the intensity of negative emotions, repetitive thinking, loss of thought control, and the strength of negative affect. The total score, which is derived by summing up the scores of all items, indicates the overall level of the measured construct.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University

IPD SHARING:
Plan to Share IPD: No